CLINICAL TRIAL: NCT00211289
Title: Trial of Education and Compliance in Heart Dysfunction. A Study Measuring the Impact of Multi-disciplinary Education as an Intervention to Increase Patient Concordance and the Cost Effectiveness of Treatment in Patients With Heart Dysfunction
Brief Title: Trial of Education and Compliance in Heart Dysfunction (TEACH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 09091E; HSFO NA-5047
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2005-06

CONDITIONS: Heart Failure
Keywords: Educational Interventions; Heart Failure; Compliance
MeSH Terms: conditions — Heart Failure; Patient Compliance

INTERVENTIONS:
Behavioral: Education by community pharmacist

SUMMARY:
The emphasis of this grant is to investigate ways to educate patients, not only to improve their knowledge about medications and diet that are important for better outcomes in heart failure, but also to try to understand how patients' beliefs about medication and diet affect their behaviour and to what extent the investigators can help patients change.

Hypotheses: Heart failure patients who receive an enhanced educational intervention from their community pharmacist will:

1. have an absolute risk reduction in the number of events of 20%,
2. be more compliant,
3. demonstrate less health-related quality of life (HRQoL) impairment as measured by disease-specific and generic HRQoL instruments and
4. have lower costs/quality adjusted life years due to fewer total events per patient.

DETAILED DESCRIPTION:
INTRODUCTION: Heart Failure (HF) is one of the leading causes of hospitalization in Canada. While great advances have been made in the treatment of this disease, factors limiting the effectiveness of treatment include: poor compliance to dietary guidelines and medications, patients' lack of understanding about the impact of their disease, a lack of understanding of the impact of their lifestyle habits on their disease and the lack of systematic monitoring of patients following hospitalization. The objective of this trial of education and compliance in heart failure patients (TEACH) is to measure in patients with heart failure who are hospitalized and then discharged into the community, the impact of a comprehensive outpatient educational intervention on:

1. a composite endpoint of mortality, readmissions and visits to the emergency room for all causes,
2. the impact of the intervention on health-related quality of life,
3. the impact of the intervention on compliance to medication and
4. the economic impact of providing such an intervention to patients. A unique component of this study is the participation of community pharmacists as part of a seamless care model and the economic and qualitative evaluation of the educational interventions.

RESEARCH DESIGN: This is a prospective, randomized controlled clinical trial in patients who are admitted to the hospital with a diagnosis of heart failure. Patients are stratified by reason for admission to the hospital. Stratum 1 includes patients whose primary reason for admission is HF and stratum 2 includes patients whose primary reason for hospital admission is not HF. The randomization will follow a cluster randomization design such that the community pharmacies will be randomized to deliver either an intervention (INTERVENTION) or usual care (CONTROL). Patients will be assigned to one of the two arms contingent upon which pharmacy they obtain most of their medications from. All patients receive standardized in-hospital education that has been previously validated (Eur J of HF, in press 2003). This education consists of educational booklets and videos on HF, health promotion and dietary information as well as relevant intervention from their community pharmacist that is aimed at helping the patients become more compliant with their medication and provide a framework of understanding that helps persistence.

HYPOTHESIS: HF patients who receive an enhanced educational intervention from their community pharmacist will:

1. have an absolute risk reduction in the number of events of 20%,
2. be more compliant,
3. demonstrate less health-related quality of life (HRQoL) impairment as measured by disease-specific and generic HRQoL instruments and
4. lower costs/quality adjusted life years (QALY) due to fewer total events per patient.

OUTCOMES: Outcomes are collected every 3 months from baseline to end of one year. Events are tracked using a comprehensive database that we have developed and validated. Further utilization data will be provided by ICES data linkage facilities and patient interviews at the time of outcome assessment. In order to measure compliance we will continue to use electronic measures known as Track Caps (MEMS). The other indirect measure is pharmacy refill data that is provided to us from all community pharmacies the patient uses. This data will be interpreted using a validated formula developed by Steiner et al. (1996). Resource use and clinical outcomes are also collected.

IMPORTANCE: Medication used to treat HF and other chronic diseases can only work, if used. We are providing a validated education intervention to patients through an existing community infrastructure with an aim to reduce morbidity and mortality and have a positive impact on HRQoL within a cost-effective framework.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of dyspnea
* Concurrent physical exam consistent with rales, S3, elevated JVP, pedal oedema
* Heart failure (HF) confirmed by attending physician, if patient is assessed by house staff
* Left ventricular ejection fraction (LVEF) < 40% on echocardiogram, nuclear scan or contrast ventriculography
* Indications for chronic medical treatment for HF
* Able and willing to give informed consent
* Over 18 years of age
* Live within London, Ontario and surrounding area, defined by the boundaries as the London and District Pharmacists' Association

Exclusion Criteria:

* Planned surgical correction for HF within 12 months
* Cor pulmonale and only right ventricular failure
* Chronic renal failure on dialysis (these patients are followed by nephrology educators)
* Other illnesses with survival anticipated for < 12 months
* Dementia documented by attending physician
* Psychiatric illness that makes it impossible to respond to education through the community pharmacist
* Planned discharge to long term institution
* Barrier to teaching (English is not the first language AND caregiver cannot provide translation to the patient to elicit the patient's responses)
* Severe alcohol or drug abuse
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Estimated)
Dates: Start 2002-07; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes: data collected on all cause mortality, all cause readmissions and all cause emergency room visits | at one year

SECONDARY OUTCOMES:
Baseline outcome measurements and quality of life | One year
Medication compliance | One year

CONTACTS AND LOCATIONS:
Overall Officials: Femida H Gwadry-Sridhar, PhD, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Hotel Dieu Grace Hospital, Windsor, Ontario